CLINICAL TRIAL: NCT01502098
Title: Effect of Postoperative Immobilization on Healing After Rotator Cuff Arthroscopic Repair With Double Row Technique in Small or Medium Ruptures. Prospective, Comparative and Randomized.
Brief Title: Effect of Postoperative Immobilization on Healing After Rotator Cuff Arthroscopic Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, Lopez Ovenza Juan Manuel, Principal Investigator, Hospital Italiano de Buenos Aires
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEPI:1780
Record Dates: First submitted 2011-12-24; First posted 2011-12-30 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2012-01

CONDITIONS: Rotator Cuff Tear
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Suburethral Slings

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early passive motion (Active Comparator): Pendulum exercises starting on the first postoperative day. The patients are instructed to commence passive range-of-motion exercises in the plane of the scapula with the assistance with the contralateral limb. Active motion exercises were not permitted until four weeks after surgery.
  Interventions: Procedure: Postoperative early passive motion
- Immobilization (No Intervention): Immobilization with sling during a month. Pendulum exercises starting on the fourth postoperative week. The patients are instructed to commence passive range-of-motion exercises in the plane of the scapula with the assistance with the contralateral limb. Active motion exercises.
  Interventions: Other: Sling

INTERVENTIONS:
Procedure: Postoperative early passive motion — Shoulder exercises starting on the first postoperative day
  Arms: Early passive motion
Other: Sling — Sling for 4 weeks
  Arms: Immobilization

SUMMARY:
The study aims to establish whether one month postoperative immobilization compared early passive motion after rotator cuff arthroscopic repair in small or medium ruptures with double row technique has any healing significance.

ELIGIBILITY:
Inclusion Criteria:

* Patients skeletally mature (older 18 years old)
* Small or medium rupture of rotator cuff
* Repaired with arthroscopic double row technique

Exclusion Criteria:

* Impossibility to perform MRI (claustrophobic, pacemaker, heart or brain metallic implants)
* AC arthritis with mumford procedure
* Smokers
* Diabetes
* Postoperative complication (severe pain, thrombosis, infection)
* Psychiatric disorder

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-06 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
MRI | 6 months

SECONDARY OUTCOMES:
ASES (American Shoulder and Elbow Surgeons Subjective Shoulder Scale) | 1, 3, 6 months
  The ASES is 100-point standardized shoulder-assessment self-report form, 50 points of which are derived from patient self-report of pain on a visual analog scale and 50 points of which are computed from a formula using the cumulative score of 10 activities of daily living derived using a four-point ordinal scale.
Range of Motion | 1, 3, 6 months
VAS of pain | 1, 3, 6 months
  visual analogue scale of pain
WORC | 1, 3, 6 months
  The Western Ontario Rotator Cuff Index (WORC) is a self-report questionnaire developed specifically to evaluate disability in persons with pathology of the rotator cuff of the shoulder.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina